# MUSIC VS MIDAZOLAM DURING PREOPERATIVE NERVE BLOCK PLACEMENT: A PROSPECTIVE, RANDOMIZED CONTROLLED STUDY

Principal Investigator Veena Graff MD

Department of Anesthesiology & Critical Care

Penn Pain Medicine Center, Tuttleman Center - Second Floor,

1840 South Street, Philadelphia, PA 19146

(570) 730-1350

Sub Investigator Nabil M Elkassabany MD

Department of Anesthesiology & Critical Care

Study Product Research selected music

IRB Number 826754

Initial version [01/12/2017] Amended [2/13/2017] Amended 12/18/2017

# **Table of Contents**

| В | ACKGR | OUND AND STUDY RATIONALE | 5 |
|---|---|---|---|
| 1 | INTR | ODUCTION | 5 |
| | 1.1 | BACKGROUND AND RELEVANT LITERATURE | 6 |
| 2 | STU | OY OBJECTIVES | 6 |
| | 2.1<br>2.2 | PRIMARY OBJECTIVESECONDARY OBJECTIVES (IF APPLICABLE) | |
| 3 | INVE | STIGATIONAL PLAN | 7 |
| | 3.1 | GENERAL DESIGN | |
| | 3.2 | ALLOCATION TO INTERVENTIONAL GROUP [IF APPLICABLE] | |
| | 3.3<br>3.4 | STUDY MEASURES | |
| | 3.4.1 | | |
| | 3.4.2 | • • | |
| 4 | STU | DY POPULATION AND DURATION OF PARTICIPATION | |
| | 4.1 | DURATION OF STUDY PARTICIPATION | |
| | 4.2 | TOTAL NUMBER OF SUBJECTS AND SITES | g |
| | 4.3 | Inclusion Criteria | |
| | 4.4 | EXCLUSION CRITERIA | |
| | 4.5<br>4.6 | SUBJECT RECRUITMENT | |
| 5 | | DY PROCEDURES | |
| J | | | |
| | 5.1 | SCREENING | |
| | 5.2 | STUDY INTERVENTION OR OBSERVATIONAL PHASE (GIVE THIS SEC | FERRORI ROCKMARK NOT DEFINED |
| | 5.2.1 | , | |
| | 5.2.2 | | |
| | 5.2.3 | Visit 3 | |
| | 5.2.4 | \ | |
| | 5.2.5 | | |
| | 5.3<br>5.4 | UNSCHEDULED VISITS | |
| | 5.4<br>5.4.1 | | |
| | 5.5 | EARLY TERMINATION VISITS | |
| | 5.6 | EFFICACY EVALUATIONS (ONLY IF APPLICABLE) | |
| | 5.7 | PHARMACOKINETIC EVALUATION (ONLY IF APPLICABLE) | |
| | 5.8 | GENETIC TESTING (ONLY IF APPLICABLE) | |
| | 5.9 | SAFETY EVALUATION (ONLY IF APPLICABLE) | |
| 6 | STA | TISTICAL PLAN | 11 |
| | 6.1 | SAMPLE SIZE AND POWER DETERMINATION | |
| | 6.2 | STATISTICAL METHODS | |
| | 6.3 | CONTROL OF BIAS AND CONFOUNDING (IF APPLICABLE, TYPICAL | |
| | 6.3.1 | IZATION IS NOT TAKING PLACE) | |
| | 6.3.2 | | |
| | 6.3.3 | | |
| | 6.3.4 | | |
| 7 | SAF | ETY AND ADVERSE EVENTS | 11 |
| | 7.1 | DEFINITIONS | 11 |
| | 7.1.1 | | |

| | 7.1.2 | Serious Adv | verse Event | t | | | | | | 12 |
|---|---|---|---|---|---|---|---|---|---|---|
| | 7.2 | RECORDING OF | ADVERSE E | EVENTS | S | | | | | 12 |
| | 7.3 | RELATIONSHIP | | | | | | | | |
| 7.4 REPORTING OF SERIOUS ADVERSE EVENTS AND UNANTI | | | | | | | | | | |
| | 7.4.1 | Follow-up F | Report | | | | | | | 12 |
| | 7.4.2 | | reporting: | notifyii | ng the stu | dy sponsor | (if applicabl | e) <b>Error! B</b> | ookmark | not |
| | <b>defi</b> i<br>7.4.3 | | afety Monit | oring F | Plan | | | | | 12 |
| 8 | STU | DY ADMINISTI | RATION, D | ATA H | ANDLIN | G AND REG | CORD KEE | PING | | 13 |
| | 8.1 | CONFIDENTIALI | TY | | | | | | | 13 |
| | 8.2 | DATA COLLECT | | | | | | | | |
| | 8.3 | RECORDS RETI | ENTION | | | | | | | 13 |
| 9 | STU | DY MONITORI | NG, AUDIT | ING, A | AND INSI | PECTING | | | | 13 |
| | 9.1 | STUDY MONITO | RING PLAN. | | | | | | | 13 |
| | 9.2 | AUDITING AND I | NSPECTING | | | | | | | 13 |
| 10 | ETH | ICAL CONSIDI | ERATIONS | | | | | | | 13 |
| | 10.1 | RISKS | | | | | | | | 13 |
| | 10.2 | BENEFITS | | | | | | | | 14 |
| | 10.3 | RISK BENEFIT A | | | | | | | | |
| | 10.4 | INFORMED CON | | | | | | | | |
| | | | | - 1 0 | | / ! ! | - I I - : £ I | : - - \ | Daakmark | |
| | 10.4. | | ns to Typica | ai Cons | sent Proc | ess (only inc | сіиае іт аррі | icable) <b>Error!</b> | DOOKIIIAIK | not |
| | 10.4.<br><b>defi</b> i | | ns to Typica | ai Cons | sent Proc | ess (only inc | сіиае іт аррі | icable) <b>Error</b> ! | DOUKIIIAIK | not |
| 11 | defii | ned.<br>DY FINANCES | | | | | | | | 14 |
| 11 | defii | ned. DY FINANCES FUNDING SOUR | | | | | | | | <b>14</b><br>14 |
| 11 | defin<br>STU<br>11.1<br>11.2 | ned. DY FINANCES FUNDING SOUR CONFLICT OF IN | CE | | | | | | | <b>14</b><br>14<br>14 |
| 11 | defin<br>STU<br>11.1<br>11.2<br>11.3 | ned. DY FINANCES FUNDING SOUR CONFLICT OF IN SUBJECT STIPE | CEVTEREST | YMENTS | <br>3 | | | | | 14<br>14<br>14<br>14 |
| 12 | defin<br>STU<br>11.1<br>11.2<br>11.3 | THE SUBJECT STIPE THE SUBJECT STIPE LICATION PLA | RCE<br>NTEREST<br>ENDS OR PAY | YMENTS | S | | ERROR! | BOOKMARK | NOT DEFI | 14<br>14<br>14<br>14<br>NED. |
| | defin<br>STU<br>11.1<br>11.2<br>11.3<br>PUB<br>REF | THE STATE OF THE S | RCE<br>NTEREST<br>NDS OR PAY | YMENTS | S | | ERROR! | BOOKMARK | NOT DEFII | 14<br>14<br>14<br>14<br>NED. |
| 12 | defin<br>STU<br>11.1<br>11.2<br>11.3<br>PUB<br>REF | THE THE PROPERTY OF THE PROPE | NTEREST | YMENTS | S | | ERROR! | BOOKMARK | NOT DEFI | 14<br>14<br>14<br>NED.<br>14<br>NED. |
| 12 | defin<br>STU<br>11.1<br>11.2<br>11.3<br>PUB<br>REF | THE STATE OF THE S | NTEREST | YMENTS | S | | ERROR! | BOOKMARK | NOT DEFI | 14<br>14<br>14<br>NED.<br>14<br>NED. |
| 12<br>13 | defin<br>STU<br>11.1<br>11.2<br>11.3<br>PUB<br>REF | THE THE PROPERTY OF THE PROPE | RCE<br>VTEREST<br>ENDS OR PAY | YMENTS | S | | ERROR!<br>ERROR! | BOOKMARK<br>BOOKMARK<br>BOOKMARK | NOT DEFII | 14<br>14<br>14<br>NED.<br>14<br>NED.<br>NED. |
| 12<br>13 | define STU 11.1 11.2 11.3 PUB REF | THE STUDIES INVOLES FUNDING SOUR CONFLICT OF IN SUBJECT STIPE LICATION PLA ERENCES ENDICES EXAMPLE: TA STUDIES INVOL | RCE<br>NTEREST<br>NDS OR PAY<br>AN | YMENTS | of Study | PROCEDURE | ERROR!<br>ERROR!<br>ERROR! | BOOKMARK BOOKMARK BOOKMARK RROR! BOOKMARK | NOT DEFII NOT DEFII NOT DEFII | 14<br>14<br>14<br>NED.<br>14<br>NED.<br>NED. |
| 12<br>13 | defin<br>STU<br>11.1<br>11.2<br>11.3<br>PUB<br>REF<br>ATT<br>APP | FUNDING SOUR CONFLICT OF IN SUBJECT STIPE LICATION PLA ERENCES ACHMENTS EXAMPLE: TA STUDIES INVOL | RCERCE | YMENTS | of Study | PROCEDURE | ERRORI ERRORI ERRORI ES E | BOOKMARK BOOKMARK BOOKMARK RROR! BOOKMARK RROR! BOOKMARK | NOT DEFII<br>NOT DEFII<br>NOT DEFII<br>ARK NOT DEF<br>ARK NOT DEF | 14 14 14 NED 14 NED. NED. SINED. SINED. |
| 12<br>13 | defin<br>STU<br>11.1<br>11.2<br>11.3<br>PUB<br>REF<br>ATT<br>APP<br>15.1<br>15.2<br>15.3<br>15.4 | FUNDING SOUR CONFLICT OF IN SUBJECT STIPE LICATION PLA ERENCES ACHMENTS ENDICES INVOL STUDIES INVOL STUDIES INVOL | RCE<br>NTEREST<br>NDS OR PAY<br>AN<br>BLE 1: SCHE<br>VING RESEA<br>VING RESEA | YMENTS | of Study<br>IRIS<br>ADIATION.<br>T SCANS. | Procedure | ERRORI ERRORI ERRORI ES EI EI EI EI EI | BOOKMARK BOOKMARK BOOKMARK RROR! BOOKMARROR! | NOT DEFII<br>NOT DEFII<br>NOT DEFII<br>ARK NOT DEF<br>ARK NOT DEF<br>ARK NOT DEF | 14 14 14 NED 14 NED. NED. SINED. SINED. SINED. SINED. SINED. |
| 12<br>13 | defin<br>STU<br>11.1<br>11.2<br>11.3<br>PUB<br>REF<br>ATT<br>APP<br>15.1<br>15.2<br>15.3<br>15.4<br>15.5 | FUNDING SOUR CONFLICT OF IN SUBJECT STIPE LICATION PLA ERENCES ACHMENTS ENDICES INVOL STUDIES INVOL STUDIES INVOL | RCE<br>NTEREST<br>NDS OR PAY<br>AN<br>BLE 1: SCHE<br>VING RESEA<br>VING RESEA | YMENTS | of Study<br>IRIS<br>ADIATION.<br>T SCANS. | Procedure | ERRORI ERRORI ERRORI ES EI EI EI EI EI | BOOKMARK BOOKMARK BOOKMARK RROR! BOOKMARROR! | NOT DEFII<br>NOT DEFII<br>NOT DEFII<br>ARK NOT DEF<br>ARK NOT DEF<br>ARK NOT DEF | 14 14 14 NED 14 NED. NED. SINED. SINED. SINED. SINED. SINED. |
| 12<br>13 | defin<br>STU<br>11.1<br>11.2<br>11.3<br>PUB<br>REF<br>ATT<br>APP<br>15.1<br>15.2<br>15.3<br>15.4<br>15.5<br>NOT DEF | FUNDING SOUR CONFLICT OF IN SUBJECT STIPE LICATION PLATERING S | RCE ENDS OR PAY AN BLE 1: SCHE VING RESEA VING RESEA VING RUCLE | EDULE ARCH MARCH CEAR ME | of Study IRIS ADIATION. T SCANS. DICINE RE | Procedure | ERROR! ERROR! ES EF EF EF SEARCH PRO | BOOKMARK BOOKMARK ROR! BOOKMARROR! BOOKMAR | NOT DEFII<br>NOT DEFII<br>ARK NOT DEF<br>ARK NOT DEF<br>ARK NOT DEF<br>ARK NOT DEF<br>OR! BOOK | 14 14 14 NED. NED. NED. SINED. SINED. SINED. SINED. MARK |
| 12<br>13 | ### defin STU ### 11.1 ### 11.2 ### 11.3 ### PUB ### REF ### ATT ### 15.1 ### 15.2 ### 15.3 ### 15.4 ### 15.5 ### NOT DEF ### Error! | FUNDING SOUR CONFLICT OF IN SUBJECT STIPE LICATION PLA ERENCES ACHMENTS EXAMPLE: TA STUDIES INVOL FINED. Reference | RCE ENDS OR PAY AN BLE 1: SCHE VING RESEA VING RESEA VING RESEA VING NUCLE SOURCE | EDULE ARCH MARCH CEAR ME | OF STUDY IRIS T SCANS. DICINE RE | Procedure | ERRORI ERRORI ERRORI ES EI EI EI EI EI | BOOKMARK BOOKMARK BOOKMARK RROR! BOOKMARROR! | NOT DEFII<br>NOT DEFII<br>NOT DEFII<br>ARK NOT DEF<br>ARK NOT DEF<br>ARK NOT DEF | 14 14 14 NED 14 NED. NED. SINED. SINED. SINED. SINED. |
| 12<br>13 | ### defin | FUNDING SOUR CONFLICT OF IN SUBJECT STIPE LICATION PLATERINGS | ANBLE 1: SCHE VING RESEA VING RESEA VING RUCLE SOURCE | EDULE ARCH MARCH CEAR ME | OF STUDY IRIS T SCANS. DICINE RE found. 20 | PROCEDURE | ERROR! ERROR! ES EF EF EF SEARCH PRO | BOOKMARK BOOKMARK ROR! BOOKMARROR! BOOKMAR | NOT DEFII NOT DEFII NOT DEFII ARK NOT DEF OR! BOOK | 14 14 14 NED 14 NED. NED. SINED. SINED. SINED. MARK NOT |
| 12<br>13 | ### defin | FUNDING SOUR CONFLICT OF IN SUBJECT STIPE LICATION PLA ERENCES ACHMENTS EXAMPLE: TA STUDIES INVOL FINED. Reference | ANBLE 1: SCHE VING RESEA VING RESEA VING NUCLE SOURCE NOT F | EDULE RACH RACH CAR ME | of Study IRIS ADIATION. T SCANS. DICINE RE found. 20 15.8SOUF | PROCEDURE | ERROR! ERROR! ES EF EF EF SEARCH PRO | BOOKMARK BOOKMARK ROR! BOOKMARROR! BOOKMAR | NOT DEFII<br>NOT DEFII<br>ARK NOT DEF<br>ARK NOT DEF<br>ARK NOT DEF<br>ARK NOT DEF<br>OR! BOOK | 14 14 14 NED 14 NED. NED. SINED. SINED. SINED. MARK NOT |

# Study Summary

| Title | MUSIC VS MIDAZOLAM DURING PREOPERATIVE NERVE BLOCK<br>PLACEMENT: A PROSPECTIVE, RANDOMIZED CONTROLLED STUDY |
|---|---|
| Short Title | Music and Preoperative Nerve Block |
| IRB Number | 826754 |
| Methodology | A prospective, randomized controlled study |
| Study Duration | One year |
| Study Center(s) | Single-center, ambulatory surgical center, at a university hospital |
| Objectives | Primary: To determine preoperative anxiety score differences between patients who receive music vs IV midazolam during preoperative nerve block placement Secondary: To evaluate differences in hemodynamics, block times, patient satisfaction scores, provider satisfaction scores, evaluation difficulty in communication between provider and patient, and adverse effects between both study groups |
| Number of Subjects | 200 |
| Main Inclusion and<br>Exclusion Criteria | Inclusion: patients who are >18 years of age who are able to give informed consent who are scheduled to receive any type of peripheral nerve block either for their primary anesthetic or for postoperative pain control in the preoperative bay at the ambulatory surgical center. Exclusion: patients who have an associated significant psychiatric disorder such as anxiety, panic disorder, depression, psychosis, or bipolar disorder; patients who are unable to give informed consent; patients who are pregnant; patients who have an underlying coagulopathy and infection, patients with hypersensitivity to midazolam, glaucoma, breastfeeding, history of renal impairment, and COPD, patient with anxiety score 50 and over. |

| | There will be two study groups who will be randomized. 1. Music group: |
|---|---|
| | patients in this group will receive research-selected music after the golden |
| | moment has been completed between the patient, provider, and nursing staff. |
| | 2. Midazolam group: patients in this group will receive IV midazolam (0.5mg to |
| | 2mg max) after the golden moment has been completed. |
| Intervention | |
| | In our daily practice, it is the provider's preference to give patients medication |
| | for sedation while conducting the preoperative nerve block. Patients do not |
| | routinely get sedation medication during the preoperative nerve block |
| | placement. |
| Statistical | |
| Methodology | 1:1 Randomized controlled study |
| Wethodology | |
| | The PI, Dr. Graff and her MD collaborator Dr. Nabil Elkassabany will be |
| | responsible for data safety and monitoring. All data will be kept in a locked |
| Data and Safety | cabinet in the MD collaborator's office. The PI and collaborators will perform |
| Monitoring Plan | safety reviews after 25 subjects are enrolled. Any protocol-related problem or |
| | deviation will be reported to Dr. Graff and/or Dr. Nabil Elkassabany as soon as |
| | possible. |

# **Background and Study Rationale**

# 1 Introduction

This document is a research protocol and the described study will be conducted in compliance with the provisions set forth in the protocol as well as, Good Clinical Practice standards, associated federal regulations, and all applicable University research requirements.

Patients often feel a tremendous amount of anxiety prior to their planned surgical procedure and anesthetic. As a result, this can affect their perioperative period by elevating their stress markers, causing various fluctuations in their hemodynamics, and poorly impacting their postoperative recovery<sup>1</sup>. A significant number of patients have anxiety about the anticipation in their overall outcome and postoperative pain control.<sup>2,3</sup>In addition to this, an increase in preoperative anxiety can result in an increase in intraoperative anesthetic requirements.<sup>3</sup> To treat preoperative anxiety, pharmacologic agents such as short-acting benzodiazepines and opioids are used as needed depending on an individual basis; however, there are known significant side effects from these medications such as respiratory depression, vital sign abnormalities, and possible apnea which limit the use of these medications and in some instances, prevent the use for preoperative anxiety. In addition to this, utilization of these medications for conscious sedation also require continuous monitoring of a patient by either anesthesia personnel or nursing staff.

Music is a non-pharmacologic intervention that has been shown to significantly decrease preoperative anxiety. This intervention can be used as an adjunct or even replace pharmacologic agents to help with preoperative anxiety. A Music is a modality that is virtually harm-free and relatively cheap in cost. Patients who are unable to tolerate pharmacologic agents to treat preoperative anxiety can greatly benefit from non-pharmacologic options such as music.

Music vs Midaz Sedation Version: 2.0

In this study, we aim to evaluate the use of music as a preoperative anxiolytic prior to the administration of a peripheral nerve block. This study will be conducted at an ambulatory surgical center in a university setting.

# 1.1 Background and Relevant Literature

Patients often feel a tremendous amount of anxiety prior to their planned surgical procedure and anesthetic. As a result, this can affect their perioperative period by elevating their stress markers, causing various fluctuations in their hemodynamics, and poorly impacting their postoperative recovery<sup>1</sup>. A significant number of patients have anxiety about the anticipation in their overall outcome and postoperative pain control<sup>2,3</sup>. In addition to this, an increase in preoperative anxiety can result in an increase in intraoperative anesthetic requirements<sup>3</sup>. To treat preoperative anxiety, pharmacologic agents such as short-acting benzodiazepines and opioids are used as needed depending on an individual basis; however, there are known significant side effects from these medications such as respiratory depression, vital sign abnormalities, and possible apnea which limit the use of these medications and in some instances, prevent the use for preoperative anxiety. In addition to this, utilization of these medications for conscious sedation also require continuous monitoring of a patient by either anesthesia personnel or nursing staff.

Music is a non-pharmacologic intervention that has been shown to significantly decrease preoperative anxiety. This intervention can be used as an adjunct or even replace pharmacologic agents to help with preoperative anxiety¹. Music is a modality that is virtually harm-free and relatively cheap in cost. Patients who are unable to tolerate pharmacologic agents to treat preoperative anxiety can greatly benefit from non-pharmacologic options such as music.

The Speilberger's validated tool, the State Trait Anxiety Inventory (STAI), is one of the best measured tools to evaluate preoperative anxiety. The STAI has been referred to as the "gold standard" in properly evaluating preoperative anxiety<sup>3</sup>. There are two components to this tool; a state portion which evaluates the current state of anxiety a patient has in a clinical setting, and a trait portion which evaluates how the patient generally feels unrelated to the clinical setting. Each of these sections have 20 items to answer and approximately takes 10-15 minutes to complete. In preoperative anxiety testing, the STAI-S is commonly used in research to properly evaluate the level of preoperative anxiety in the current clinical setting. Marteau and her colleagues have developed a shortened STAI version, the STAI-6, that has also been validated <sup>5</sup>. The shortened STAI-6 tool has six questions and may be more beneficial to use in a high turnover, ambulatory surgical center setting as it only takes a few minutes to complete.

We will be using the STAI-6 short form questionnaire to score the preoperative anxiety levels in our patient population.

# 2 Study Objectives

# 2.1 Primary Objective

To determine preoperative anxiety score differences between patients who receive music vs IV midazolam during their preoperative nerve block placement.

# 2.2 Secondary Objectives (if applicable)

To evaluate differences in hemodynamics, block times, patient satisfaction scores, provider satisfaction scores, evaluation difficulty in communication between provider and patient, and adverse effects between both study groups

# 3 Investigational Plan

# 3.1 General Design

This will be a prospective, randomized controlled study. Participants will be randomized to receiving research-selected music versus IV midazolam (0.5mg to 2mg max) during their preoperative peripheral nerve block placement.

# 3.2 Allocation to Interventional Group [if applicable]

Subjects will be randomized to either music or IV midazolam. Subjects will be randomized in a one to one fashion and the randomization will take place using a computer-generated algorithm.

# 3.3 Study Measures

There will be two study groups who will be randomized. 1. Music group: patients in this group will receive research-selected music after the golden moment has been completed between the patient, provider, and nursing staff. 2. Midazolam group: patients in this group will receive IV midazolam (0.5mg to 2mg max) after the golden moment has been completed.

A pre-anxiety score will be obtained using the STAI-6 validated tool after the patient has signed the informed consent. After the golden moment is completed, the intervention will start. Once the nerve block is completed, a post anxiety score will be obtained using STAI-6 validated tool. The post anxiety score will be obtained from the start of the anxiolytic intervention in both groups.

For our primary outcome measure, we will use the short form of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI-6) to measure pre procedure and post procedure anxiety levels (see below). The shortened STAI-6 tool has six questions and may be more beneficial to use in a high turnover, ambulatory surgical center setting as it only takes a few minutes to complete. In the original 20-item STAI-State tool, the scores range from 20 to 80. A score greater than 50 on the original 20-item scale is associated with a high level of anxiety. The population normal score is approximately 35 (Speilberger 1983). In the STAI-6 tool, there are six questions with a Likert scale from 1 to 4. This gives a score range from 6 to 24. To create scores compatible with the original STAI-S scores, the STAI-6 scores will be divided by 6 and multiplied by 20 to give a range from 20 to 80.

# Appendix A: Self-evaluation questionnaire (Y-6 item)

| Name Date |
|---|
| A number of statements which people have used to describe themselves are given below. Read each statement and then |
| circle the most appropriate number to the right of the statement to indicate how you feel right now, at this moment. |
| There are no right or wrong answers. Do not spend too much time on any one statement but give the answer which |
| seems to describe your present feelings best. |

| | Not at all | Somewhat | Moderately | Very much |
|---|---|---|---|---|
| 1, I feel calm | 1 | 2 | 3 | 4 |
| 2. I am tense | 1 | 2 | 3 | 4 |
| <ol><li>I feel upset</li></ol> | 1 | 2 | 3 | 4 |
| 4. I am relaxed | 1 | 2 | 3 | 4 |
| <ol><li>I feel content</li></ol> | 1 | 2 | 3 | 4 |
| <ol><li>I am worried</li></ol> | 1 | 2 | 3 | 4 |

Please make sure that you have answered all the questions.

For our secondary outcome measure, we will obtain the following information:

1. Patient satisfaction scores using a 10-point visual analogue scale (VAS) as follows:

"Using any number from 0 to 10, where 0 is the <u>WORST</u> experience possible and 10 is the <u>BEST</u> experience possible, what number would you use to rate your overall preoperative experience while getting a peripheral nerve block placed?"



2. Provider satisfaction scores using a 10-point visual analogue scale (VAS) as follows:

"Using any number from 0 to 10, where 0 is the <u>WORST</u> experience possible and 10 is the <u>BEST</u> experience possible, what number would you use to rate your overall preoperative experience while placing a peripheral nerve block for your patient?"



3. Evaluation of communication difficulties between provider and patient by asking one question on a 5-point Likert scale:

From provider to patient:

"I found it difficult to communicate with the patient while doing the preoperative nerve block."

- A. Strongly Disagree
- B. Disagree
- C. Neutral
- D. Agree
- E. Strongly Agree

From patient to provider:

- "I found it difficult to communicate with the physician while the preoperative nerve block was being done on me."
  - A. Strongly Disagree
  - B. Disagree
  - C. Neutral
  - D. Agree
  - E. Strongly Agree

# 3.4 Study Endpoints

# 3.4.1 Primary Study Endpoint

The primary end point will be to determine differences in the preoperative anxiety scores using the STAI-6 tool between the music group and the IV midazolam group.

Music vs Midaz Sedation Version: 2.0

# 3.4.2 Secondary Study Endpoints

The secondary end points will be to determine any differences in patient satisfaction scores, provider satisfaction scores, evaluation of difficulties in communication between provider and patient, hemodynamics, block times, and adverse effects including paresthesia's, patchy block, failed block, and serious adverse effects including bleeding, infection, paralysis, local anesthetic systemic toxicity between both groups.

# 4 Study Population and Duration of Participation

The study population will include patients who are >18 years of age, who will give informed consent in receiving a peripheral nerve block in the preoperative bay for their primary anesthetic and/or for their postoperative pain control.

We will exclude the following: patients who have an associated significant psychiatric disorder such as anxiety, panic disorder, depression, psychosis, or bipolar disorder; patients who are unable to give informed consent; patients who are pregnant; patients who have an underlying coagulopathy and infection.

# 4.1 Duration of Study Participation

The study duration will be from the time informed consent occurs to after the perioperative block has been completed; after the start of the anxiolytic intervention (music vs IV midazolam). Once the post-anxiety STAI-6 score has been obtained, the study is complete.

# 4.2 Total Number of Subjects and Sites

Total number of subjects will be 200; 100 in the music group and 100 in the IV midazolam group. Study will take place at Penn Medicine University City, PMUC.

#### 4.3 Inclusion Criteria

Patients who are >18 years of age, who will give informed consent in receiving a peripheral nerve block in the preoperative bay for their primary anesthetic and/or for their postoperative pain control.

# 4.4 Exclusion Criteria

We will exclude the following: patients who have an associated significant psychiatric disorder such as anxiety, panic disorder, depression, psychosis, or bipolar disorder; patients who are unable to give informed consent; patients who are pregnant; patients who have an underlying coagulopathy and infection, patients with hypersensitivity to midazolam, glaucoma, breastfeeding, history of renal impairment, and COPD, patient with anxiety score 50 and over.

# 4.5 Subject Recruitment

All patients will be screened initially either at the preoperative surgical clinic visit or prior to the day of surgery via telephone once they are scheduled for surgery. Any patient that cannot be reached will be approached in the preoperative bay during the preoperative period of their planned surgery. Subjects will be given the details about the study and given adequate time to read the consent form and talk the study over with family that accompanies them.

# 4.6 Vulnerable Populations:

Children, pregnant women, fetuses, neonates, or prisoners are not included in this research study.

# 5 Study Procedures

# 5.1 Screening

The general flow of the study will be conducted as follows:

- Research coordinator will call or approach patients who are scheduled for a surgical
  procedure that is planning for a peripheral nerve block either for the primary anesthetic or for
  postoperative pain control to be placed in the preoperative bay in the ambulatory surgical
  center.
- Research coordinator will discuss the purpose of our study and explain the study in detail for the patient. If a patient agrees to participate, then we will have the patient sign the informed consent for the study. If patient is on the phone and decides to participate, the patient will sign the informed consent upon arriving to PMUC.

# 5.1.1 Visit

- Once the patient signs the informed consent for the peripheral nerve block by anesthesia team. The patient randomized will be revealed to either music or IV midazolam. The preprocedure anxiety score will then be obtained using the STAI-6 validated tool.
- 4. The golden moment will be conducted between the patient, provider, and nursing staff. Once this golden moment is completed, the anxiolytic intervention will start (music or IV midazolam)\*
- 5. The preoperative nerve block will be conducted by the regional anesthesia block team.
- 6. Once the nerve block is complete, we will obtain the post-procedure anxiety score using the STAI-6 validated tool.
- 7. Once the post-procedure anxiety score has been obtained, we will also obtain the patient satisfaction score, the provider satisfaction score, and the evaluation of any difficulties in communication between the provider and patient. After these questions have been obtained, the study is complete.

\*Research selected music will be provided for the patient via headphones. When providing music in the preoperative period for patients to obtain the anxiolytic benefit (Bradt 2013). There is however limited data on utilizing music in the preoperative data while conducting a procedure.

Patients do not routinely get sedation medication while undergoing a preoperative peripheral nerve block. Sedation medication is administered based on provider preference. This decision is made on a case by case basis. If sedation medication is used, IV midazolam is the common medication used. The IV midazolam dosage for preoperative anxiolysis ranges from 0.5mg to 2mg max.

Peripheral nerve blocks are conducted under ultrasound guidance according to standard practice at PMUC.

Vital signs such as heart rate, blood pressure, respiratory rate, and oxygen saturation are routinely obtained as a part of standard of care if sedation medication is used and when peripheral nerve blocks are placed.

Starting block time and ending block time are routinely obtained as a part of the patient record.

During this entire process, patient demographics, hemodynamics (heart rate, blood pressure, oxygen saturation, and respiratory rate), block times (start and end time), and any adverse effects including paresthesia's, patchy block, failed block, and serious adverse effects including bleeding, infection, paralysis, local anesthetic systemic toxicity will be recorded as the routine part of practice.

Music vs Midaz Sedation Version: 2.0

# 5.2 Subject Withdrawal

Subjects may withdraw from the study at any time without impact to their care. They may also be discontinued from the study at the discretion of the Investigator for lack of adherence to intervention or study procedures or AEs. It will be documented whether or not each subject completes the study.

# 5.2.1 Data Collection and Follow-up for Withdrawn Subjects

Data will still be collected for subjects who withdrawal from the study. In cases where subjects wish to withdrawn PHI consent they will be able to do so by telling a study team member in person or through information provided on the ICF.

# 5.3 Safety Evaluation

When evaluating safety, the doctors will look at any reported AE's as well as patients who are unwilling or unable to adhere to the randomized allocation. If patients in either group have more than 25% deviation rate the inclusion and exclusion as well as block method will be reevaluated to better limit deviations.

#### 6 Statistical Plan

# 6.1 Sample Size and Power Determination

Based on a previous study by Bringman et.al. the mean (SD) of STAI anxiety score is 34(8) <sup>4</sup>. A clinically meaningful decrease, as determined by the Cochrane review group was 0.5 of SD.<sup>1,6</sup> Our sample size calculation to detect a 4-point change in pain score (p less than 0.05 significance level) was 86 patients ( $\alpha$ =0.05, power=90%). We will inflate out sample size by 15% to account for any missing data or any withdrawal from the study; therefore, our estimated sample size will be 100 patients per group.

# 6.2 Statistical Methods

Statistical analyses will be performed using STATA 13 statistical software (Dallas, TX). Demographic or other categorical data will be analyzed using T test or Fishers exact test as appropriate. Repeated measurements (STAI-6 scores) will be analyzed by using the t-test or Mann-Whitney U-test as appropriate. Normally distributed data will be presented as means ± SE of the mean (SEM), non-normally distributed data are presented as medians ± quartiles (interquartile range) and categorical data will be presented as raw data and as frequencies. The alpha level for all analyses was set as P less than 0.05.

#### 6.2.1 Baseline Data

Demographic or other categorical data will be analyzed using T test or Fishers exact test as appropriate.

# **6.2.2** Analysis of Primary Outcome of Interest

Repeated measurements (STAI-6 scores) will be analyzed by using the t-test or Mann-Whitney U-test as appropriate.

# 7 Safety and Adverse Events

This section provides the safety management plans for the study. This section should be consistent with the Penn IRB guidelines tailored to the requirements specific for each study. It should describe how safety reporting will be monitored and take place over the course of the trial.

#### 7.1 Definitions

# 7.1.1 Adverse Event

Study definition of an adverse event (AE). Can include the Penn IRB definition of an adverse event unless there are some differences in the adverse event definitions for this particular study. Standard definition of an adverse event as follows:

Music vs Midaz Sedation Version: 2.0

An adverse event (AE) is any symptom, sign, illness or experience that develops or worsens in severity during the course of the study. Intercurrent illnesses or injuries should be regarded as adverse events. Abnormal results of diagnostic procedures are considered to be adverse events if the abnormality:

- results in study withdrawal
- is associated with a serious adverse event
- is associated with clinical signs or symptoms
- leads to additional treatment or to further diagnostic tests
- is considered by the investigator to be of clinical significance

#### 7.1.2 Serious Adverse Event

#### Serious Adverse Event

Adverse events are classified as serious or non-serious. A serious adverse event is any AE that is:

- fatal
- life-threatening
- requires or prolongs hospital stay
- results in persistent or significant disability or incapacity
- required intervention to prevent permanent impairment or damage
- a congenital anomaly or birth defect
- an important medical event

# 7.2 Recording of Adverse Events

Information on all adverse events will be recorded immediately in the source document, and also in the appropriate adverse event module of the case report form (CRF). All clearly related signs, symptoms, procedures results will be recorded in the source document.

All adverse events occurring during the study period will be recorded. The clinical course of each event will be followed until resolution, stabilization, or until it has been determined that the study intervention or participation is not the cause. Serious adverse events that are still ongoing at the end of the study period will be followed up to determine the final outcome. Any serious adverse event that occurs after the study period and is considered to be possibly related to the study intervention or study participation will be recorded and reported.

# 7.3 Relationship of AE to Study

The PI will supervise the assessment of relationship of each adverse even to the study procedures. The adverse events, if such occurs, will be classified as definitely related, probably related, possibly related, unlikely or unrelated.

# 7.4 Reporting of Adverse Events and Unanticipated Problems

The Investigator will promptly notify the Penn IRB of all on-site unanticipated, Adverse Events that are related to the research activity. Other unanticipated problems related to the research involving risk to subjects or others will also be reported promptly. Written reports will be filed using the HS-ERA and in accordance with the Penn IRB timeline of 10 working days.

# 7.4.1 Follow-up Report

If an AE has not resolved at the time of the initial report and new information arises that changes the investigator's assessment of the event, a follow-up report including all relevant new or reassessed information (e.g., concomitant medication, medical history) should be submitted to the IRB. The investigator is responsible for ensuring that all SAEs are followed until either resolved or stable.

# 7.4.2 Data and Safety Monitoring Plan

The PI, Dr. Graff and her collaborator Dr. Nabil Elkassabany will be responsible for data safety and monitoring. All paper data will be kept in a locked cabinet in the MD collaborator's office. The PI and

Music vs Midaz Sedation Version: 2.0

collaborators will perform safety reviews after 25 patients are enrolled. Any protocol-related problem or deviation will be reported to Dr. Graff and/or Dr. Nabil Elkassabany as soon as possible.

# 8 Study Administration, Data Handling and Record Keeping

# 8.1 Confidentiality

Information about study subjects will be kept confidential and managed according to the requirements of the Health Insurance Portability and Accountability Act of 1996 (HIPAA). Those regulations require a signed subject authorization informing the subject of the following:

- What protected health information (PHI) will be collected from subjects in this study
- Who will have access to that information and why
- Who will use or disclose that information
- The rights of a research subject to revoke their authorization for use of their PHI.

In the event that a subject revokes authorization to collect or use PHI, the investigator, by regulation, retains the ability to use all information collected prior to the revocation of subject Study date will be stored on a Penn institutionally secured and managed server specific to the Anesthesiology Department in a locked folder only for this protocol.

# 8.2 Data Collection and Management

Demographic information will be collected from patient charts. Information about sedation onset, block start and stop as well as survey information will be captured on paper that will be stored on Penn campus in secured building in locked office in locked filing cabinets. Subjects will be given a study number at time of enrollment. De-identified data will be inputted into a department and folder password secured excel sheet.

Once study analysis is complete identifiable information linking subject to study number will be destroyed/ deleted.

# 8.3 Records Retention

Records will be retained up to 3 years after the completion of research. Electronic records of directly collected data will subsequently be destroyed from electronic server.

# 9 Study Monitoring, Auditing, and Inspecting

# 9.1 Study Monitoring Plan

The study will be monitored by Dr. Graff and Dr. Elkassabany.

# 9.2 Auditing and Inspecting

The investigator will permit study-related monitoring, audits, and inspections by the IRB, government regulatory bodies, and University compliance and quality assurance groups of all study related documents (e.g. source documents, regulatory documents, data collection instruments, study data etc.). The investigator will ensure the capability for inspections of applicable study-related facilities.

#### 10 Ethical Considerations

Study will be submitted to the Penn IRB for approval before study enrollment begins. Any changes to the protocol will we preapproved by the IRB before any changes to study practice is made.

# 10.1 Risks

The risks of the study are related to the administration of midazolam which include tenderness and pain during injection at IV site. This risk is addressed in the local block consent form and thus is not putting subjects at a greater risk.

Music vs Midaz Sedation Version: 2.0

#### 10.2 Benefits

The individual subjects may not receive any benefit from participating in this study. Potential benefit could be increased relaxation and lower anxiety from music sedation or midazolam. For the study population this study hopes to prove that non medicinal sedation is adequate for subject comfort and a decrease in anesthetics can be achieved.

#### 10.3 Risk Benefit Assessment

The potential benefits are greater to the limited risks for patients thus this study should be conducted.

# 10.4 Informed Consent Process / HIPAA Authorization

All subjects for this study will be provided a consent form describing this study providing sufficient information for subjects to make an informed decision about their participation in this study. This consent form will be submitted with the protocol for review and approval by the IRB for the study. The formal consent of a subject, using the IRB-approved consent form, must be obtained before that subject undergoes any study procedure. The subject, must sign the consent form, and the investigator-designated research professional obtaining the consent. Subjects will be consented by the study Principal Investigator, or appropriate designee, in perioperative holding room assigned at check in. Potential subjects will review the consent form in detail with the person designated to consent (either PI or CRC) and have the ability to review consent with family or friends that accompanied them to PMUC.

# 11 Study Finances

# 11.1 Funding Source

This study is not funded.

#### 11.2 Conflict of Interest

No conflicts of interest have been noted by initial study team if conflict arises the IRB will be notified according to regulations. All University of Pennsylvania Investigators will follow the University of Pennsylvania Policy on Conflicts of Interest Related to Research.

# 11.3 Subject Stipends or Payments

Subjects will not be paid for study.

# 12 References

- 1. Bradt J, Dileo C, Shim M. Music interventions for preoperative anxiety. *The Cochrane database of systematic reviews*. 2013(6):Cd006908.
- 2. Kain ZN, Sevarino F, Alexander GM, Pincus S, Mayes LC. Preoperative anxiety and postoperative pain in women undergoing hysterectomy. A repeated-measures design. *Journal of psychosomatic research*. 2000;49(6):417-422.
- 3. Maranets I, Kain ZN. Preoperative anxiety and intraoperative anesthetic requirements. *Anesthesia and analgesia*. 1999;89(6):1346-1351.
- 4. Bringman H, Giesecke K, Thorne A, Bringman S. Relaxing music as pre-medication before surgery: a randomised controlled trial. *Acta anaesthesiologica Scandinavica*. 2009;53(6):759-764.
- 5. Marteau TM, Bekker H. The development of a six-item short-form of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI). *The British journal of clinical psychology*. 1992;31 ( Pt 3):301-306.
- 6. Sloan JA. Assessing the minimally clinically significant difference: scientific considerations, challenges and solutions. *Copd.* 2005;2(1):57-62.